CLINICAL TRIAL: NCT02784756
Title: Cell-Mediated Immunity Based Primary Prophylaxis for CMV Infection in Organ Transplant Recipients: A Multi-Center Study
Brief Title: Cell-Mediated Immunity Based Primary Prophylaxis for CMV Infection in Organ Transplant Recipients
Acronym: QFT-CMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian National Transplant Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-9877
Record Dates: First submitted 2016-02-10; First posted 2016-05-27 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cytomegalovirus Viraemia
Keywords: Quantiferon-CMV; solid organ transplant; CMV Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quantiferon-CMV assay (Other): All patients will receive a CMV-immunity test at specific time points during the study. This is a single arm design
  Interventions: Device: Quantiferon-CMV assay

INTERVENTIONS:
Device: Quantiferon-CMV assay

SUMMARY:
The study will prospectively determine the clinical utility of CMV cell-mediated immunity using the Quantiferon test. The investigators will use the assay results to tailor the duration of CMV prophylaxis in solid organ transplant patients.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) disease is an important cause of morbidity in solid organ transplantation recipients and remains the most common opportunistic viral infection in these patients. Standard CMV prevention strategies include universal prophylaxis and pre-emptive therapy with viral load monitoring. However, neither of these strategies has been successful in eliminating CMV disease as seen by high rates of viremia, incidence, and CMV recurrence despite treatment. Recently, the Quantiferon-CMV assay has been shown to predict late CMV reactivation after prophylaxis and to be predictive of viral progression and the need for antiviral therapy in organ transplant recipients who develop low level CMV viremia. The purpose of the current study is to test the clinical strategy of using the Quantiferon-CMV assay in guiding the duration of primary CMV prophylaxis in solid organ transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney, kidney-pancreas, liver transplant recipient, or heart transplant recipient
* CMV D+/R- patient or any R+ patient who received antithymocyte globulin induction therapy

Exclusion Criteria:

* Unable to comply with protocol
* Campath (Alemtuzumab) induction
* Receiving another investigational compound for CMV treatment or prophylaxis.
* Allergy to valganciclovir or ganciclovir
* Receiving an investigational compound for prevention or treatment of rejection, or participating in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-06; Primary Completion 2020-02 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Symptomatic CMV disease | 1 year
  Number of participants with symptomatic CMV disease (including viral syndrome and tissue invasive disease) at 1 year post-transplant.

SECONDARY OUTCOMES:
Occurrence of CMV viremia | 1 year
  Occurrence of CMV viremia as measured by QuantiFERON-CMV assay (> 1000 IU/mL)
positive vs. negative cell-mediated immunity assays | 1 year
  Incidence of positive vs. negative cell-mediated immunity assays post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Atul Humar, MD, Principal Investigator — University Health Network, Toronto; Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (6):
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Paul's Hospital - Providence Health, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibson L. An Interferon-gamma Release Assay for Evaluation of Cell-mediated Immunity in Infants With Congenital Cytomegalovirus Infection. Clin Infect Dis. 2021 Aug 2;73(3):374-375. doi: 10.1093/cid/ciaa700. No abstract available. PMID 32504089